CLINICAL TRIAL: NCT04828824
Title: Reduction of Premature Discontinuation of Contraceptive Implants by Advance Provision of an OCP-based Participant Intervention: Randomized Clinical Trial
Brief Title: Premature Discontinuation of Contraceptive Implants
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-2750
Record Dates: First submitted 2021-03-30; First posted 2021-04-02 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Contraception Behavior
MeSH Terms: conditions — Contraception Behavior | interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- COCR Arm (Experimental): Participants in the COCR arm will receive three packs of combined oral contraceptive pills (35mcg ethinyl estradiol/norgestimate) and a specific protocol for their use for bothersome bleeding.
  Interventions: Drug: Ethinyl Estradiol / Norgestimate Oral Tablet
- SOC Arm (No Intervention): Participants in the SC arm will be offered care according to our standardized protocol, which may include STI testing, reassurance and monitoring, prescription of COCs if desired, or removal.

INTERVENTIONS:
Drug: Ethinyl Estradiol / Norgestimate Oral Tablet — Those who desire COCs as an intervention are prescribed (over the phone) or given (in person) 3 packs of COCs. They are told to take one pill per day until the first pack is complete and save the remaining 2 packs for possible future use.
  Arms: COCR Arm

SUMMARY:
To compare rates of etonogestrel implant discontinuation in implant initiators who are given advance provision of combined oral contraceptive pills (COCs) and a bleeding rescue regimen (COCR intervention) to participants given standard counseling (comparator).

DETAILED DESCRIPTION:
Objective:

To compare rates of etonogestrel implant discontinuation in implant initiators who are given advance provision of combined oral contraceptive pills (COCs) and a bleeding rescue regimen (COCR intervention) to participants given standard counseling (comparator).

Secondary Objectives:

To determine if participants initiating the contraceptive implant who are also provided COCR are more likely than participants receiving standard counseling to:

1. report higher levels of satisfaction with their contraceptive implant at one year following initiation
2. require less clinical follow-up and clinical resources in the year following initiation.

ELIGIBILITY:
Inclusion Criteria:

1. You are between ages of 14 to 22.9 years.
2. Started etonogestrel implant for the first time and have never used the implant before.

Exclusion Criteria:

1. There is any contraindication to estrogen containing birth control.
2. Desire of pregnancy in next 12 months.
3. Plans to move from the area in next 12 months and is not able to come to the clinic.

Ages: 14 Years to 23 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant Continuation | 12 months post-insertion
  We will assess continuation of use of the contraceptive implant.

SECONDARY OUTCOMES:
Satisfaction with contraceptive implant | 3, 6, and 12 months post-insertion
  We will assess satisfaction with bleeding profile and overall satisfaction using a Likert scale ("very satisfied", "somewhat satisfied" and "not satisfied").

OTHER OUTCOMES:
Implant-related health care interactions | within 12 months of insertion
  We will assess the number of healthcare interactions (phone calls, visits, messages, prescription refills) that are related to the use of the contraceptive implant or oral contraceptives dispensed in this study using the electronic medical record system.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided